CLINICAL TRIAL: NCT00159588
Title: Medication-overuse Headache (MOH): Withdrawal or Use of Preventative Medications Directly? A Randomized Multi-centre Follow-up.
Brief Title: Medication-overuse Headache (MOH): Withdrawal or Use of Preventative Medications Directly?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004/534; NCT00159588
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Results first posted 2021-12-01 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2021-12

CONDITIONS: Headache
Keywords: Medication-overuse headache; preventative medication; controls; follow-up; randomized; abrupt withdrawal
MeSH Terms: conditions — Headache; Headache Disorders, Secondary | interventions — Angiotensin Receptor Antagonists; Valproic Acid; Antidepressive Agents, Tricyclic; Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Prophylaxis from the start (Active Comparator): Use of preventive drugs from the start without abrupt withdrawal
  Interventions: Drug: Betablockers or other preventive drugs based on primary headache type
- Abrupt withdrawal (Other): Device: Abrupt withdrawal. Standard out-patients detoxication program including telephone call after 2 weeks and rescue medicine up to 2 days/week
  Interventions: Drug: Betablockers or other preventive drugs based on primary headache type
- Controls (Other): Active control: No instruction for abrupt withdrawal or prophylactic treatment. The controls finished the study period after 5 months observation, and were then offered the optimal type of treatment
  Interventions: Drug: Betablockers or other preventive drugs based on primary headache type

INTERVENTIONS:
Drug: Betablockers or other preventive drugs based on primary headache type — Several preventive drugs based on each individual regarding type of original headache type (i.e angiotensin II blockers, betablockers, valproate, tricyclic antidepressants or gabapentin)
  Other Names: angiotensin II blockers, betablockers, valproate, tricyclic antidepressants or gabapentin

SUMMARY:
It is a common belief that patients with MOH rarely respond of preventative medications whilst overusing acute medications. However, no randomized trial has been done previously to prove such statement. Based on some clinical experiences, our hypothesis are patients with probably MOH may benefit from use of preventive medications better than treatment with abrupt withdrawal or no specific treatment.

DETAILED DESCRIPTION:
This randomized multi-centre study started January 2004, and patients with probably MOH have been included from five different University hospitals in Norway. The last patient was included November 9th 2006, final inclusion date was December 31th 2006. At this time a total of 64 patients with probable MOH according to the International Classification of Headache Disorders, 2nd Edition (2004) were included.

The included patients were randomized to one out of three possible options:

1. Abrupt withdrawal of the acute medication(s) they have been overusing. After 3 month: use of preventative medication (best choice)in those who need such treatment, 12 month follow-up.
2. Start with preventative medication (best choice) directly without abrupt withdrawal, 12 month follow-up.
3. No specific treatment (controls), 5 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* fulfill 8.2.7 probably medication-overuse headache according to the International Classification of Headache Disorders, 2th Edition (2004)

Exclusion Criteria:

* No benefit of all available preventative medications
* no benefit of abrupt withdrawal lasting more than 3 weeks of acute medication that has been overused
* cluster headache
* chronic paroxysmal hemicrania
* hemicrania continua, pregnancy
* use of pain killers for other reasons than headache
* other reasons for chronic daily headache than medication-overuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2004-01; Primary Completion 2006-11 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Knut Hagen, MD; PhD,, Study Chair — Dept. of Neurology, St. Olavs University Hospital, Trondheim, Norway
Locations (1):
- Knut Hagen, Trondheim, Norway

REFERENCES:
- [Result] Hagen K, Albretsen C, Vilming ST, Salvesen R, Gronning M, Helde G, Gravdahl G, Zwart JA, Stovner LJ. Management of medication overuse headache: 1-year randomized multicentre open-label trial. Cephalalgia. 2009 Feb;29(2):221-32. doi: 10.1111/j.1468-2982.2008.01711.x. Epub 2008 Sep 24. PMID 18823363
- [Result] Hagen K, Stovner LJ. A randomized controlled trial on medication-overuse headache: outcome after 1 and 4 years. Acta Neurol Scand Suppl. 2011;(191):38-43. doi: 10.1111/j.1600-0404.2011.01542.x. PMID 21711255

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 64 randomized, 3 excluded not fulfilling the inclusion criteria after the baseline period
Groups:
- Preventive Drugs From the Start: Use of preventive drugs from the start without abrupt withdrawal. This group was not explicitly advised to withdraw overused medication. Preventive medication was started on day 1, based on a priority list of medicines (Betablockers, candesartan, topiramate, amitriptyline or other preventive relevant drugs. For each patient preventive agent was chosen on the basis of a list of specifications considering the primary headache, side-effects of the drug and what they have tried before.
- Abrupt Withdrawal: Device: Abrupt withdrawal
- Controls: Active control: No instruction for abrupt withdrawal or prophylactic treatment
Period: 5 Month Follow-up
Arm/Group | Preventive Drugs From the Start | Abrupt Withdrawal | Controls
Started | 19 | 22 | 20
Completed (Fulfilled the 5-month visit) | 17 | 18 | 18
Not Completed | 2 | 4 | 2
Not completed — Withdrawal by Subject | 2 | 4 | 2
Period: 1-year Follow-up for Group 1 and 2
Arm/Group | Preventive Drugs From the Start | Abrupt Withdrawal | Controls
Started | 17 | 18 | 18
Completed | 16 | 14 | 18
Not Completed | 1 | 4 | 0

BASELINE CHARACTERISTICS:
Population: Three out of 64 randomized patients were excluded because they had <15 headache days/months at baseline. Baseline data was available in 61 who meet the inclusion criteria.
Groups:
- Preventive Drugs From the Start: Preventive medication started day 1 without explicit advice of withdrawal of overused medication
- Abrupt Withdrawal: Standard out-patient detoxication program
- Controls: Did not get a new preventive medication or direct advice to stop use of analgesics
- Total: Total of all reporting groups
Arm/Group | Preventive Drugs From the Start | Abrupt Withdrawal | Controls | Total
Number analyzed (Participants) | 19 | 22 | 20 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 22 | 20 | 61
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (10) | 42.1 (9) | 38.7 (11) | 40.9 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 11 | 36
  Male | 8 | 8 | 9 | 25

OUTCOME MEASURES:

1. Primary Outcome: Headache Days
Description: Change in Headache days per month
Time Frame: 5 month
Population: Headache diary information available
Measure: Median (95% Confidence Interval); unit: days/month
Arm/Group | Prophylaxis From the Start | Abrupt Withdrawal | Controls
Number analyzed (Participants) | 17 | 18 | 18
days/month | 7.2 [2.7 to 11.8] | 4.2 [3.3 to 7.4] | 1.6 [0.1 to 1.8]
Statistical Analysis 1: Comparison: Prophylaxis From the Start vs Abrupt Withdrawal vs Controls; Kruskal-Wallis test; Test type: Superiority; p = 0.056, Kruskal-Wallis — Between-group analysis

2. Secondary Outcome: Headache Index
Description: Headache index (HI) per month calculated by the sum of products of headache days /month combined with mean daily hours with headache and mean daily headache severity on days with headache. High HI reflect high headache burden
Time Frame: 5-month follow-up
Population: Headache diary information available
Measure: Mean (95% Confidence Interval); unit: headache index per month
Groups:
- Preventive Drugs From the Start: Use of preventive drugs from the start without abrupt withdrawal
  Betablockers or other preventive drugs: Several preventive drugs based on each individual
Arm/Group | Preventive Drugs From the Start | Abrupt Withdrawal | Controls
Number analyzed (Participants) | 17 | 18 | 18
headache index per month | 169 [89 to 248] | 371 [296 to 513] | 302 [252 to 424]
Statistical Analysis 1: Comparison: Preventive Drugs From the Start vs Abrupt Withdrawal vs Controls; Kruskal-Wallis test; Test type: Superiority — Between-group analysis; p = 0.012, t-test, 2 sided — Between-group analysis; Kruskal-Wallis test

ADVERSE EVENTS:
Time Frame: 5 months for controls, 1 year for the other two groups
Description: Adverse events collected in the case report form (CRF) during consultation at 1, 3 and 5 months and during the 12-month follow up visit
Arm/Group | Preventive Drugs From the Start | Abrupt Withdrawal | Controls
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 1/17 | 3/20 | 1/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preventive Drugs From the Start (N=17) | Abrupt Withdrawal (N=20) | Controls (N=19)
dizziness (Ear and labyrinth disorders) | 1 (1) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes